CLINICAL TRIAL: NCT03069989
Title: A Study of Single Doses to Evaluate the Safety, Tolerability, Pharmacokinetics and Target Engagement of Nebulised GSK3008348 in Idiopathic Pulmonary Fibrosis Patients, Using Positron Emission Tomography (PET) Imaging
Brief Title: Single Doses of GSK3008348 in Idiopathic Pulmonary Fibrosis (IPF) Participants Using Positron Emission Tomography (PET) Imaging
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sufficient information was gathered from cohort 1 to terminate the study without proceeding to optional cohort 2.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204715; 2016-003674-41 (EudraCT Number)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Tolerability; IPF; PET imaging; Idiopathic Pulmonary Fibrosis; Safety; Pharmacokinetics; Double-blind
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — GSK3008348

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 GSK3008348 (Experimental): Participants will receive a single nebulized dose of GSK3008348 during each of 2 planned dosing periods and up to 3 microdose administrations of [18F]-FBA-A20FMDV2 for the PET scanning in period 2.
  Interventions: Drug: GSK3008348; Drug: [18F]-FBA-A20FMDV2
- Cohort 1 Placebo (Placebo Comparator): Participants will receive a single nebulized dose of placebo during each of 2 planned dosing periods and up to 3 microdose of [18F]-FBA-A20FMDV2 for the PET scanning in period 2.
  Interventions: Drug: Placebo; Drug: [18F]-FBA-A20FMDV2
- Cohort 2 GSK3008348 (Experimental): Participants will receive a single nebulized dose of GSK3008348 during each of 2 planned dosing periods and up to 3 microdose administrations of [18F]-FBA-A20FMDV2 for the PET scanning in period 2.
  Interventions: Drug: GSK3008348; Drug: [18F]-FBA-A20FMDV2
- Cohort 2 Placebo (Placebo Comparator): Participants will receive a single nebulized dose of placebo during each of 2 planned dosing periods and up to 3 microdose of [18F]-FBA-A20FMDV2 for the PET scanning in period 2.
  Interventions: Drug: Placebo; Drug: [18F]-FBA-A20FMDV2

INTERVENTIONS:
Drug: GSK3008348 — Solution for nebulisation. Available as clear colorless to pale yellow colored solution in a 5mL vial with 20 millimeter (mm) stopper and aluminium seal yellow colored solution in a 5mL vial with 20 millimeter (mm) stopper and aluminium seal.
  Arms: Cohort 1 GSK3008348; Cohort 2 GSK3008348
Drug: Placebo — Solution for nebulisation. Available as clear colorless to pale yellow colored solution in a 5mL vial with 20mm stopper and aluminium seal.
  Arms: Cohort 1 Placebo; Cohort 2 Placebo
Drug: [18F]-FBA-A20FMDV2 — Radio-labeled peptide ligand for PET scan. Available as intravenous (IV) infusion, 20 mL.

SUMMARY:
GSK3008348 is being developed as a treatment for IPF. A first-time-in-human study showed that single nebulized doses of 1-3000 micrograms (mcg) GSK3008348 in healthy volunteers were well tolerated, with pharmacokinetic (PK) exposures within the defined limits set in the protocol. The proposed study is a 2-cohort study of single doses, intended to evaluate the safety, tolerability and PK of the drug in participants with IPF not currently treated with pirfenidone or nintedanib, and to obtain preliminary information on target engagement. Cohort 1 will be a 2-period, randomized, double-blind, placebo-controlled group with at least 7 days washout between doses, and follow-up period of up to 7-14 days. Cohort 2 is optional. It will be designed to further explore safety and to provide additional information on the target engagement profile of GSK3008348. The total duration of the study will be up to 62 days.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged >= 50 years, and female participants aged >=55 years, at the time of signing the informed consent.
* Diagnosis of definite or probable IPF as determined by a responsible and experienced chest physician and based on established criteria defined by the American Thoracic Society/European Respiratory Society Internationale Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias.
* Ambulant and capable of attending outpatient visits.
* FVC > 50 percent predicted and DLCO > 40 percent predicted.
* Body weight >= 45 kilograms (kg) and body mass index (BMI) within the range 18.0-35.0 kg/square meter (inclusive).
* Male and female
* Male participants: A male participant must agree to use contraception as detailed in this protocol during the study and for at least 90 days after the follow up visit, and refrain from donating sperm during this period.
* Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and not a woman of childbearing potential (WOCBP) as defined in the protocol.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions, listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* ALT and bilirubin > 1.5x upper limit of normal (ULN; isolated bilirubin > 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin < 35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT corrected (QTc) > 450 milliseconds (msec), or QTc > 480 msec in participants with Bundle Branch Block.
* Current IPF exacerbation, or upper or lower respiratory tract infection on admission to the clinical unit.
* History of or suffers from claustrophobia, or unable to lie flat and still on their back for up to 2 hrs in the PET scanner.
* Extent of emphysema greater than the extent of fibrotic change on High-Resolution Computed Tomography (HRCT) scan, based on investigator judgment.
* FEV1/FVC ratio < 0.70 at screening (post-bronchodilator).
* History of sensitivity to the study treatment, or components thereof, or a history of drug or other allergy that, in the opinion of the investigators or Medical Monitor, contraindicates their participation.
* Any current oro-pharygneal disease or disorders as judged by the investigator.
* Currently taking pirfenidone or nintedanib, or received pirfenidone or nintedanib within 30 days of the first dose of study treatment.
* Taken, within 7 days or 5 half-lives (whichever is longer) before the first dose of study treatment, organic anion transporter (OAT) substrates with a narrow therapeutic index (example: methotrexate and tenofovir), vitamins, or dietary or herbal supplements, unless in the opinion of the investigator and sponsor the supplement will not interfere with the study medication.
* Long-term continuous home oxygen therapy (use of oxygen that is only intermittent and for symptom relief is acceptable).
* Participation in a clinical trial and receipt of an investigational medicinal product within the following time period before the first dose in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 new investigational medicinal products within 12 months before the first dose.
* Presence of Hepatitis B surface antigen (HBsAg) at screening, or positive Hepatitis C antibody test result at screening or within 3 months before the first dose of study treatment.

Note: participants with a positive Hepatitis C antibody test because of previous, resolved disease can be enrolled if a confirmatory negative Hepatitis C Ribonucleic Acid (RNA) test is obtained.

* Previous or current exposure to animals that may harbour Food and Mouth Disease Virus (FMDV2).
* Previous long term (>= 3 months) residence in a country where FMDV2 is endemic (such as certain areas of Africa, Asia and South America.
* Where participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 56 days.
* History of drug or alcohol abuse that in the opinion of the investigator affects their participation in the study.
* Exposure to ionizing radiation in excess of 10 Millisievert (mSv) above background over the previous 3 year period as a result of occupational exposure or previous participation in research studies. Clinically justified (therapeutic or diagnostic) exposures are not included in the exposure calculation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 sites in the United Kingdom from 13-June-2017 to 18-July-2018. At the interim analysis following review of Cohort 1 data it was agreed to stop the study without proceeding into optional Cohort 2.
Pre-assignment Details: A total of 11 participants were screened, of which 3 were screening failures. Two screening failure participants did not meet inclusion/exclusion criteria and 1 participant withdrew consent. Hence, 8 participants were enrolled in this study.
Groups:
- Placebo: Participants received a single dose of placebo (solution), inhaled via nebulization on Day 1 in dosing periods 1 and 2. In dosing period 2 only, they received up to 150 MBq of a [18F]-FBA-A20FMDV2, via IV infusion, prior to PET imaging at Baseline, 30 minutes and approximately 24 hours post-GSK3008348 dose. Total [18F]-FBA-A20FMDV2 administration was <=100 mcg per participant. A wash out period of at least 7 and no more than 28 days was maintained between doses in Periods 1 and 2.
- GSK3008348 1000 mcg: Participants received a single dose of GSK3008348 1000 mcg (solution), inhaled via nebulization on Day 1 in dosing periods 1 and 2. In dosing period 2 only, they received up to 150 MBq of [18F]-FBA-A20FMDV2, via IV infusion, prior to PET imaging at Baseline, 30 minutes and approximately 24 hours post-GSK3008348 dose. Total [18F]-FBA-A20FMDV administration was <=100 mcg per participant. A wash out period of at least 7 and no more than 28 days was maintained between doses in Periods 1 and 2.
Period: Dosing Period 1 (Up to 2 Days)
Arm/Group | Placebo | GSK3008348 1000 mcg
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0
Period: Wash Out Period (Up to 28 Days))
Arm/Group | Placebo | GSK3008348 1000 mcg
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0
Period: Dosing Period 2 (Up to 16 Days)
Arm/Group | Placebo | GSK3008348 1000 mcg
Started | 3 | 5
Completed | 2 | 5
Not Completed | 1 | 0
Not completed — Protocol-defined stop criteria reached | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3008348 1000 mcg | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.3 (3.06) | 73.6 (2.30) | 72.4 (2.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Period 2: Volume of Distribution (VT) of [18F]-FBA-A20FMDV2 in the Whole Lung (Not Corrected for Air Volume) at 30 Minutes Post-dose Compared to Pre-dose
Description: The change in the uptake of [18F]-FBA-A20FMDV2 in the whole lung, assessed by VT derived from kinetic analysis of the dynamic PET data, was used to evaluate target engagement in the lung after single nebulized doses of GSK3008348. The per-Protocol population consisted of all participants in the Intent-to-Treat population who comply with the protocol and that had at least one evaluable PET measurement post-dose.
Time Frame: Baseline (pre-dose) and 30 minutes post-dose
Population: Per-Protocol Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per cubic centimeter(mL/cm^3)
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Milliliter per cubic centimeter(mL/cm^3)
  Baseline | 1.664 (19.67) | 1.503 (37.32)
  30 minutes post-dose PET scan 1 | 1.572 (8.56) | 1.198 (44.37)

2. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician. Intent-to-Treat population consisted of all randomized participants who received at least one dose of study treatment.
Time Frame: Up to 62 days
Population: Intent-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Participants
  AEs | 1 | 3
  SAEs | 0 | 0

3. Primary Outcome: Period 1: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count and White Blood Cell (WBC) Count
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet count, platelet count and WBC count. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Giga cells per liter
  Basophils | 0.000 (0.0000) | -0.008 (0.0179)
  Eosinophils | 0.000 (0.0000) | 0.018 (0.0402)
  Lymphocytes | 0.267 (0.0577) | -0.086 (0.3361)
  Monocytes | -0.033 (0.0577) | -0.106 (0.1232)
  Total neutrophils | 0.300 (0.5292) | -0.762 (0.8135)
  Platelet count | -3.0 (16.46) | -24.2 (11.69)
  WBC count | 0.467 (0.4933) | -0.982 (0.9509)

4. Primary Outcome: Period 2: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count and WBC Count
Description: as for outcome 3
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Giga cells per liter
  Basophils | 0.010 (0.0424) | -0.034 (0.0365)
  Eosinophils | 0.025 (0.0071) | -0.030 (0.1051)
  Lymphocytes | 0.485 (0.1061) | 0.168 (0.3269)
  Monocytes | -0.050 (0.1414) | -0.046 (0.1172)
  Total neutrophils | -0.155 (0.5728) | -0.866 (0.6179)
  Platelet count | -2.5 (16.26) | 15.8 (12.87)
  WBC count | 0.270 (0.5657) | -0.748 (0.7351)

5. Primary Outcome: Period 1: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Grams per liter | -4.3 (2.89) | -4.4 (6.84)

6. Primary Outcome: Period 2: Change From Baseline in Hematology Parameter: Hemoglobin
Description: as for outcome 5
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Grams per liter | -4.0 (5.66) | -8.8 (3.56)

7. Primary Outcome: Period 1: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Proportion of red blood cells in blood | 0.000 (0.0000) | -0.016 (0.0270)

8. Primary Outcome: Period 2: Change From Baseline in Hematology Parameter: Hematocrit
Description: as for outcome 7
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Proportion of red blood cells in blood | -0.013 (0.0057) | -0.028 (0.0141)

9. Primary Outcome: Period 1: Change From Baseline in Hematology Parameter: Mean Corpuscle Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: mean corpuscle hemoglobin. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Picrograms
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Picrograms | -0.30 (0.265) | 0.10 (0.500)

10. Primary Outcome: Period 2: Change From Baseline in Hematology Parameter: Mean Corpuscle Hemoglobin
Description: as for outcome 9
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picrograms
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Picrograms | -0.75 (0.212) | -0.50 (0.361)

11. Primary Outcome: Period 1: Change From Baseline in Hematology Parameter: Mean Corpuscle Volume
Description: Blood samples were collected to analyze the hematology parameter: mean corpuscle volume. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Femtoliters | 1.00 (1.000) | -0.58 (1.559)

12. Primary Outcome: Period 2: Change From Baseline in Hematology Parameter: Mean Corpuscle Volume
Description: as for outcome 11
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Femtoliters | -2.35 (1.061) | -1.62 (1.213)

13. Primary Outcome: Period 1: Change From Baseline in Hematology Parameter: Red Blood Cell Count
Description: Blood samples were collected to analyze the hematology parameter: red blood cell count. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Trillion cells per liter | -0.093 (0.0702) | -0.168 (0.2946)

14. Primary Outcome: Period 2: Change From Baseline in Hematology Parameter: Red Blood Cell Count
Description: as for outcome 13
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Trillion cells per liter | -0.010 (0.1556) | -0.226 (0.1372)

15. Primary Outcome: Period 1: Change From Baseline in Chemistry Parameters: Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Creatine Kinase and Gamma Glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: alkaline phosphatase, alanine amino transferase, aspartate amino transferase, creatine kinase and gamma glutamyl transferase. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population. Only those participants available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
International units per liter
  Alkaline phosphatase, n=3,5 | -1.7 (1.53) | -3.4 (10.43)
  Alanine amino transferase, n=3,5 | 1.3 (1.53) | -0.6 (1.14)
  Aspartate amino transferase, n=2,3: number analyzed (Participants) | 2 | 3
  Aspartate amino transferase, n=2,3 | 0.0 (2.83) | -0.3 (3.06)
  Creatine kinase, n=3,5 | -95.0 (76.62) | -13.8 (9.31)
  Gamma glutamyl transferase, n=3,5 | -1.0 (1.00) | -1.2 (2.17)

16. Primary Outcome: Period 2: Change From Baseline in Chemistry Parameters: Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Creatine Kinase and Gamma Glutamyl Transferase
Description: as for outcome 15
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
International units per liter
  Alkaline phosphatase, n=2,4: number analyzed (Participants) | 2 | 4
  Alkaline phosphatase, n=2,4 | -4.5 (0.71) | -14.5 (17.41)
  Alanine amino transferase, n=2,4: number analyzed (Participants) | 2 | 4
  Alanine amino transferase, n=2,4 | 4.0 (1.41) | -0.5 (3.70)
  Aspartate amino transferase, n=2,2: number analyzed (Participants) | 2 | 2
  Aspartate amino transferase, n=2,2 | 2.5 (2.12) | -6.5 (6.36)
  Creatine kinase, n=2,4: number analyzed (Participants) | 2 | 4
  Creatine kinase, n=2,4 | -94.0 (127.28) | -7.8 (20.45)
  Gamma glutamyl transferase, n=2,3: number analyzed (Participants) | 2 | 3
  Gamma glutamyl transferase, n=2,3 | -5.0 (1.41) | -4.0 (2.65)

17. Primary Outcome: Period 1: Change From Baseline in Chemistry Parameters: Albumin and Total Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin and total protein. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Grams per liter
  Albumin | -1.3 (1.15) | -2.6 (3.78)
  Total protein | -1.7 (2.89) | -4.0 (6.40)

18. Primary Outcome: Period 2: Change From Baseline in Chemistry Parameters: Albumin and Total Protein
Description: as for outcome 17
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Grams per liter
  Albumin | 1.5 (0.71) | -1.4 (1.52)
  Total protein | -0.5 (0.71) | -7.4 (5.55)

19. Primary Outcome: Period 1: Change From Baseline in Chemistry Parameters: Direct Bilirubin, Total Bilirubin and Creatinine
Description: Blood samples were collected to analyze the chemistry parameters: direct bilirubin, total bilirubin and creatinine. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Micromoles per liter
  Direct bilirubin, n=2,4: number analyzed (Participants) | 2 | 4
  Direct bilirubin, n=2,4 | 0.0 (0.00) | -0.5 (1.73)
  Total bilirubin, n=3,5 | -3.0 (1.00) | -2.2 (6.46)
  Creatinine, n=3,5 | -6.0 (15.10) | -3.6 (5.59)

20. Primary Outcome: Period 2: Change From Baseline in Chemistry Parameters: Direct Bilirubin, Total Bilirubin and Creatinine
Description: as for outcome 19
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population. Only those participants with available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Micromoles per liter
  Direct bilirubin, n=1,3: number analyzed (Participants) | 1 | 3
  Direct bilirubin, n=1,3 | 2.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed. | 1.3 (1.53)
  Total bilirubin, n=2,5: number analyzed (Participants) | 2 | 5
  Total bilirubin, n=2,5 | -2.5 (0.71) | -4.8 (4.02)
  Creatinine, n=2,5: number analyzed (Participants) | 2 | 5
  Creatinine, n=2,5 | -5.0 (16.97) | -2.0 (5.61)

21. Primary Outcome: Period 1: Change From Baseline in Chemistry Parameters: Calcium, Glucose, Potassium, Sodium and Blood Urea Nitrogen
Description: Blood samples were collected to analyze the chemistry parameters: calcium, glucose, potassium, sodium and blood urea nitrogen. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Millimoles per liter
  Calcium, n=3,5 | -0.103 (0.0961) | -0.024 (0.1097)
  Glucose, n=3,5 | 1.17 (1.858) | 1.06 (1.126)
  Potassium, n=2,5: number analyzed (Participants) | 2 | 5
  Potassium, n=2,5 | -0.10 (0.000) | -0.48 (0.311)
  Sodium, n=3,5 | -2.7 (1.15) | -0.2 (1.64)
  Blood urea nitrogen, n=3,5 | -0.27 (1.234) | 0.14 (1.174)

22. Primary Outcome: Period 2: Change From Baseline in Chemistry Parameters: Calcium, Glucose, Potassium, Sodium and Blood Urea Nitrogen
Description: as for outcome 21
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Millimoles per liter
  Calcium, n=2,5 | -0.125 (0.0778) | -0.158 (0.1033)
  Glucose, n=2,5 | -0.25 (0.778) | -1.06 (1.403)
  Potassium, n=2,4: number analyzed (Participants) | 2 | 4
  Potassium, n=2,4 | 0.00 (0.141) | -0.20 (0.583)
  Sodium, n=2,5 | 0.5 (2.12) | 0.4 (3.36)
  Blood urea nitrogen, n=2,5 | -0.25 (0.354) | -0.06 (0.950)

23. Primary Outcome: Period 1: Number of Participants With Abnormal Urinalysis Results by Dipstick
Description: Urine samples were collected at indicated time points to analyze urinalysis parameters including specific gravity, potential of hydrogen, glucose, protein, blood and ketones by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as positive, Trace, 1+, 2+, 3+ and 4+, indicating proportional concentrations in the urine sample. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Only categories with abnormal urinalysis values are presented.
Time Frame: Baseline (Day -1) and 24 hours post-GSK3008348 dose
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Participants
  Urine occult blood- Baseline, 1+: n=3,5 | 0 | 1
  Urine occult blood- 24 hours, Trace: n=3,4: number analyzed (Participants) | 3 | 4
  Urine occult blood- 24 hours, Trace: n=3,4 | 0 | 1
  Urine occult blood- 24 hours, 1+: n=3,4: number analyzed (Participants) | 3 | 4
  Urine occult blood- 24 hours, 1+: n=3,4 | 0 | 1
  Urine protein- Baseline, 1+: n=3,4: number analyzed (Participants) | 3 | 4
  Urine protein- Baseline, 1+: n=3,4 | 1 | 0
  Urine protein - 24 hours, 1+: n=3,4: number analyzed (Participants) | 3 | 4
  Urine protein - 24 hours, 1+: n=3,4 | 0 | 1

24. Primary Outcome: Period 2: Number of Participants With Abnormal Urinalysis Results by Dipstick
Description: as for outcome 23
Time Frame: Baseline (Day -1), 24 hours post-GSK3008348 dose and Day 15 (follow-up)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Participants
  Urine occult blood- Baseline, Trace: n=2,5: number analyzed (Participants) | 2 | 5
  Urine occult blood- Baseline, Trace: n=2,5 | 0 | 1
  Urine occult blood- Day 15, Trace: n=3,5 | 0 | 1
  Urine glucose- 24 hours, 100 mg/dL : n=2,5: number analyzed (Participants) | 2 | 5
  Urine glucose- 24 hours, 100 mg/dL : n=2,5 | 0 | 1
  Urine ketones - 24 hours, 5mg/dL: n=3,4: number analyzed (Participants) | 3 | 4
  Urine ketones - 24 hours, 5mg/dL: n=3,4 | 0 | 2
  Urine proteins- Baseline, Trace: n=2,5: number analyzed (Participants) | 2 | 5
  Urine proteins- Baseline, Trace: n=2,5 | 0 | 1
  Urine proteins- 24 hours, Trace: n=2,5: number analyzed (Participants) | 2 | 5
  Urine proteins- 24 hours, Trace: n=2,5 | 0 | 1
  Urine proteins- Day 15, Trace: n=3,5 | 0 | 1

25. Primary Outcome: Period 1: Change From Baseline in Vital Signs: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: SBP and DBP were measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1), 0.5, 2, 4, 8 and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Millimeters of mercury
  DBP- 0.5 hours | 3.3 (9.29) | 2.4 (9.91)
  DBP- 2 hours | 1.3 (1.15) | -0.6 (3.21)
  DBP- 4 hours | -7.0 (5.29) | 0.2 (6.80)
  DBP- 8 hours | -0.7 (9.29) | 1.4 (10.36)
  DBP- 24 hours | -5.7 (5.51) | -4.4 (6.31)
  SBP- 0.5 hours | 16.3 (24.17) | 2.2 (20.07)
  SBP- 2 hours | 5.0 (3.61) | -11.0 (4.36)
  SBP- 4 hours | -1.7 (4.73) | -4.8 (14.75)
  SBP- 8 hours | 12.0 (23.90) | 1.8 (16.53)
  SBP- 24 hours | 1.3 (11.59) | -5.0 (12.51)

26. Primary Outcome: Period 2: Change From Baseline in Vital Signs: DBP and SBP
Description: as for outcome 25
Time Frame: Baseline (Day -1), 30 minutes (post-PET scan), Day 1 (prior to discharge) and Day 2 (pre-PET scan)
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Millimeter of mercury
  DBP-30 minutes post-PET scan | 17.0 (12.73) | 4.2 (6.91)
  DBP- Day 1 prior to discharge | 10.0 (14.14) | -3.6 (8.05)
  DBP- Day 2 pre-PET scan | 7.5 (20.51) | -4.8 (4.44)
  SBP- 30 minutes post-PET scan | 13.5 (20.51) | 7.2 (7.89)
  SBP- Day 1 prior to discharge | 10.0 (12.73) | -6.0 (12.19)
  SBP- Day 2 pre-PET scan | -3.0 (19.80) | -8.6 (16.56)

27. Primary Outcome: Period 1: Change From Baseline in Vital Signs: Heart Rate
Description: Heart rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1), 0.5, 2, 4, 8 and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Beats per minute
  0.5 hours | -0.3 (9.29) | -7.0 (11.11)
  2 hours | 4.0 (4.58) | -3.0 (10.49)
  4 hours | 12.3 (9.81) | -2.4 (6.23)
  8 hours | 17.3 (2.08) | -1.4 (10.11)
  24 hours | 6.7 (3.51) | 0.8 (5.93)

28. Primary Outcome: Period 2: Change From Baseline in Vital Signs: Heart Rate
Description: as for outcome 27
Time Frame: Baseline (Day -1), 30 minutes (post-PET scan), Day 1 (prior to discharge) and Day 2 (pre-PET scan)
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Beats per minute
  30 minutes post-PET scan | -5.5 (6.36) | -10.2 (3.77)
  Day 1 prior to discharge | 3.0 (4.24) | -5.0 (6.78)
  Day 2 pre-PET scan | -5.5 (13.44) | -9.8 (4.97)

29. Primary Outcome: Period 1: Change From Baseline in Vital Sign: Respiration Rate
Description: Respiration rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1), 0.5, 2, 4, 8 and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Breaths per minute
  0.5 hours | -0.3 (1.53) | 1.2 (2.17)
  2 hours | 1.0 (1.00) | 2.8 (3.70)
  4 hours | 1.0 (1.00) | 1.6 (2.19)
  8 hours | 0.3 (0.58) | 2.2 (3.56)
  24 hours | -0.7 (1.15) | 1.0 (2.00)

30. Primary Outcome: Period 2: Change From Baseline in Vital Sign: Respiration Rate
Description: as for outcome 29
Time Frame: Baseline (Day -1), 30 minutes (post-PET scan), Day 1 (prior to discharge) and Day 2 (pre-PET scan)
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Breaths per minute
  30 minutes post-PET scan | 0.0 (2.83) | 0.0 (0.00)
  Day 1 prior to discharge | 0.0 (2.83) | 2.8 (1.10)
  Day 2 pre-PET scan | -0.5 (0.71) | 1.0 (2.24)

31. Primary Outcome: Period 1: Change From Baseline in Vital Sign: Temperature
Description: Temperature was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1), 0.5, 2, 4, 8 and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Celsius
  0.5 hours | 0.27 (0.231) | 0.0 (0.346)
  2 hours | 0.30 (0.656) | 0.00 (0.265)
  4 hours | 0.20 (0.265) | -0.02 (0.327)
  8 hours | 0.43 (0.289) | 0.28 (0.319)
  24 hours | 0.60 (0.361) | 0.10 (0.292)

32. Primary Outcome: Period 2: Change From Baseline in Vital Sign: Temperature
Description: as for outcome 31
Time Frame: Baseline (Day -1), 30 minutes (post-PET scan), Day 1 (prior to discharge) and Day 2 (pre-PET scan)
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Celcius
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
Celcius
  30 minutes post-PET scan | -0.25 (0.919) | 0.06 (0.537)
  Day 1 prior to discharge | -0.05 (0.778) | 0.34 (0.786)
  Day 2 pre-PET scan | -0.35 (1.061) | 0.06 (0.518)

33. Primary Outcome: Period 1: Number of Participants With Abnormal Findings for 12-lead Electrocardiograms (ECG) Parameters
Description: Triplicate 12-lead ECG were obtained to measure ECG parameters. Abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS). Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Pre-dose (Day -1), 0.5, 2, 4, 8 and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Participants
  Pre-dose measurement 1, NCS | 2 | 4
  Pre-dose measurement 1, CS | 0 | 0
  Pre-dose measurement 2, NCS | 2 | 3
  Pre-dose measurement 2, CS | 0 | 0
  Pre-dose measurement 3, NCS | 3 | 3
  Pre-dose measurement 3, CS | 0 | 0
  0.5 hours measurement 1, NCS | 2 | 4
  0.5 hours measurement 1, CS | 0 | 0
  0.5 hours measurement 2, NCS | 3 | 4
  0.5 hours measurement 2, CS | 0 | 0
  0.5 hours measurement 3, NCS | 3 | 4
  0.5 hours measurement 3, CS | 0 | 0
  2 hours measurement 1, NCS | 3 | 3
  2 hours measurement 1, CS | 0 | 0
  2 hours measurement 2, NCS | 3 | 3
  2 hours measurement 2, CS | 0 | 0
  2 hours measurement 3, NCS | 3 | 3
  2 hours measurement 3, CS | 0 | 0
  4 hours measurement 1, NCS | 3 | 4
  4 hours measurement 1, CS | 0 | 0
  4 hours measurement 2, NCS | 3 | 4
  4 hours measurement 2, CS | 0 | 0
  4 hours measurement 3, NCS | 3 | 4
  4 hours measurement 3, CS | 0 | 0
  8 hours measurement 1, NCS | 3 | 4
  8 hours measurement 1, CS | 0 | 0
  8 hours measurement 2, NCS | 3 | 4
  8 hours measurement 2, CS | 0 | 0
  8 hours measurement 3, NCS | 3 | 4
  8 hours measurement 3, CS | 0 | 0
  24 hours measurement 1, NCS | 3 | 4
  24 hours measurement 1, CS | 0 | 0
  24 hours measurement 2, NCS | 3 | 4
  24 hours measurement 2, CS | 0 | 0
  24 hours measurement 3, NCS | 2 | 4
  24 hours measurement 3, CS | 0 | 0

34. Primary Outcome: Period 2: Number of Participants With Abnormal Findings for 12-lead ECG Parameters
Description: Triplicate 12-lead ECG were obtained to measure ECG parameters. Abnormal findings were categorized as CS and NCS. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Pre-dose (Day -1), 30 minutes (post-PET scan), Day 1 (prior to discharge), Day 2 (pre-PET scan) and Day 15 (follow-up)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Participants
  Pre-dose measurement 1, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  Pre-dose measurement 1, NCS,n=2,5 | 0 | 5
  Pre-dose measurement 1, CS,n=2,5: number analyzed (Participants) | 2 | 5
  Pre-dose measurement 1, CS,n=2,5 | 0 | 0
  Pre-dose measurement 2, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  Pre-dose measurement 2, NCS,n=2,5 | 0 | 5
  Pre-dose measurement 2, CS,n=2,5: number analyzed (Participants) | 2 | 5
  Pre-dose measurement 2, CS,n=2,5 | 0 | 0
  Pre-dose measurement 3, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  Pre-dose measurement 3, NCS,n=2,5 | 0 | 5
  Pre-dose measurement 3, CS,n=2,5: number analyzed (Participants) | 2 | 5
  Pre-dose measurement 3, CS,n=2,5 | 0 | 0
  30 minutes measurement 1, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  30 minutes measurement 1, NCS,n=2,5 | 1 | 4
  30 minutes measurement 1, CS,n=2,5: number analyzed (Participants) | 2 | 5
  30 minutes measurement 1, CS,n=2,5 | 0 | 0
  30 minutes measurement 2, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  30 minutes measurement 2, NCS,n=2,5 | 1 | 4
  30 minutes measurement 2, CS,n=2,5: number analyzed (Participants) | 2 | 5
  30 minutes measurement 2, CS,n=2,5 | 0 | 0
  30 minutes measurement 3, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  30 minutes measurement 3, NCS,n=2,5 | 1 | 4
  30 minutes measurement 3, CS,n=2,5: number analyzed (Participants) | 2 | 5
  30 minutes measurement 3, CS,n=2,5 | 0 | 0
  Day 1 measurement 1, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 1 measurement 1, NCS,n=2,5 | 1 | 4
  Day 1 measurement 1, CS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 1 measurement 1, CS,n=2,5 | 0 | 0
  Day 1 measurement 2, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 1 measurement 2, NCS,n=2,5 | 1 | 4
  Day 1 measurement 2, CS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 1 measurement 2, CS,n=2,5 | 0 | 0
  Day 1 measurement 3, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 1 measurement 3, NCS,n=2,5 | 1 | 4
  Day 1 measurement 3, CS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 1 measurement 3, CS,n=2,5 | 0 | 0
  Day 2 measurement 1, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 2 measurement 1, NCS,n=2,5 | 2 | 3
  Day 2 measurement 1, CS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 2 measurement 1, CS,n=2,5 | 0 | 0
  Day 2 measurement 2, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 2 measurement 2, NCS,n=2,5 | 2 | 3
  Day 2 measurement 2, CS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 2 measurement 2, CS,n=2,5 | 0 | 0
  Day 2 measurement 3, NCS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 2 measurement 3, NCS,n=2,5 | 2 | 4
  Day 2 measurement 3, CS,n=2,5: number analyzed (Participants) | 2 | 5
  Day 2 measurement 3, CS,n=2,5 | 0 | 0
  Day 15 measurement 1, NCS,n=3,5 | 1 | 3
  Day 15 measurement 1, CS,n=3,5 | 0 | 0
  Day 15 measurement 2, NCS,n=3,5 | 0 | 3
  Day 15 measurement 2, CS,n=3,5 | 0 | 0
  Day 15 measurement 3, NCS,n=3,5 | 1 | 3
  Day 15 measurement 3, CS,n=3,5 | 0 | 0

35. Primary Outcome: Period 1: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC)
Description: FEV1 and FVC is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. FEV1 and FVC was measured using standard spirometry equipment. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day -1), 1 hour and 24 hours post-GSK3008348 dose
Population: Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 3 | 5
Liters
  FEV1: 1 hour | 0.003 (0.0808) | -0.058 (0.0881)
  FEV1: 24 hours | -0.117 (0.0702) | -0.036 (0.0879)
  FVC: 1 hour | 0.067 (0.0833) | 0.086 (0.3474)
  FVC: 24 hours | -0.050 (0.1411) | -0.010 (0.1208)

36. Secondary Outcome: Period 1: Area Under the Plasma Concentration-time Curve From Zero Hours to Time (AUC[0-t]) After Single Dose Administration of GSK3008348
Description: Blood samples were collected to evaluate the pharmacokinetics of GSK3008348 at the indicated time points. The pharmacokinetic parameters were calculated by standard non-compartmental analysis. Pharmacokinetic population consisted of all participants in the Intent-To-Treat population receiving active dose for whom a pharmacokinetic sample was analyzed.
Time Frame: Pre-dose, and at 0.25, 0.5, 1, 2, 4, 8, 12, 18 and 24 hours post-GSK3008348 dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picograms per milliliter
Arm/Group | GSK3008348 1000 mcg
Number analyzed (Participants) | 5
Hours*picograms per milliliter | 64638.3 (58)

37. Secondary Outcome: Period 2: AUC(0-t) After Single Dose Administration of GSK3008348
Description: Blood samples were collected to evaluate the pharmacokinetics of GSK3008348 at the indicated time points. The pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, and at 0.25, 0.5, 2, 4, 22 and 30 hours post-GSK3008348 dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram per milliliter
Arm/Group | GSK3008348 1000 mcg
Number analyzed (Participants) | 5
Hours*picogram per milliliter | 66122.5 (44)

38. Secondary Outcome: Period 1: Area Under the Plasma Concentration-time Curve From Zero Hours to Infinity (AUC[0-infinity]) After Single Dose Administration of GSK3008348
Description: as for outcome 37
Time Frame: Pre-dose, and at 0.25, 0.5, 1, 2, 4, 8, 12, 18 and 24 hours post-GSK3008348 dose
Population: Pharmacokinetic Population. Only those participants with data available at the indicated data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picograms per milliliter
Arm/Group | GSK3008348 1000 mcg
Number analyzed (Participants) | 4
Hours*picograms per milliliter | 67715.8 (80)

39. Secondary Outcome: Period 2: AUC(0-infinity) After Single Dose Administration of GSK3008348
Description: as for outcome 37
Time Frame: Pre-dose, and at 0.25, 0.5, 2, 4, 22 and 30 hours post-GSK3008348 dose
Population: Pharmacokinetic Population. Data were not analyzed for AUC(0-infinity) as there were not enough data points collected for a terminal slope required to calculate AUC(0-infinity).
Arm/Group | GSK3008348 1000 mcg
Number analyzed (Participants) | 0

40. Secondary Outcome: Period 1: Maximum Observed Plasma Drug Concentration (Cmax) After Single Dose Administration of GSK3008348
Description: as for outcome 37
Time Frame: Pre-dose, and at 0.25, 0.5, 1, 2, 4, 8, 12, 18 and 24 hours post-GSK3008348 dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | GSK3008348 1000 mcg
Number analyzed (Participants) | 5
Picograms per milliliter | 14050.4 (38)

41. Secondary Outcome: Period 2: Cmax After Single Dose Administration of GSK3008348
Description: as for outcome 37
Time Frame: Pre-dose, and at 0.25, 0.5, 2, 4, 22 and 30 hours post-GSK3008348 dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | GSK3008348 1000 mcg
Number analyzed (Participants) | 5
Picograms per milliliter | 10418.2 (31)

42. Secondary Outcome: Period 1: Time of Occurrence of Cmax (Tmax) After Single Dose Administration of GSK3008348
Description: as for outcome 37
Time Frame: Pre-dose, and at 0.25, 0.5, 1, 2, 4, 8, 12, 18 and 24 hours post-GSK3008348 dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3008348 1000 mcg
Number analyzed (Participants) | 5
Hours | 0.50 [0.4 to 0.5]

43. Secondary Outcome: Period 2: Tmax After Single Dose Administration of GSK3008348
Description: as for outcome 37
Time Frame: Pre-dose, and at 0.25, 0.5, 2, 4, 22 and 30 hours post-GSK3008348 dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3008348 1000 mcg
Number analyzed (Participants) | 5
Hours | 0.47 [0.4 to 0.5]

44. Secondary Outcome: Period 1: Terminal Phase Half-life (t1/2) After Single Dose Administration of GSK3008348
Description: as for outcome 37
Time Frame: Pre-dose, and at 0.25, 0.5, 1, 2, 4, 8, 12, 18 and 24 hours post-GSK3008348 dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK3008348 1000 mcg
Number analyzed (Participants) | 5
Hours | 10.6 (21)

45. Secondary Outcome: Period 2: t1/2 After Single Dose Administration of GSK3008348
Description: as for outcome 37
Time Frame: Pre-dose, and at 0.25, 0.5, 2, 4, 22 and 30 hours post-GSK3008348 dose
Population: Pharmacokinetic Population. Data were not analyzed for t1/2 as there were not enough data points collected for a terminal slope required to calculate t1/2.
Arm/Group | GSK3008348 1000 mcg
Number analyzed (Participants) | 0

46. Secondary Outcome: Period 2: VT of [18F]-FBAA20FMDV2 in the Whole Lung (Not Corrected for Air Volume) Approximately 24 Hours Post-dose Compared to Pre-dose
Description: The changes in the uptake of [18F]-FBA-A20FMDV2 in the whole lung, assessed by VT derived from kinetic analysis of the dynamic PET data was used to evaluate target engagement in the lung after single nebulized doses of GSK3008348
Time Frame: Baseline (pre-dose) and 24 hours post-dose PET scan 2
Population: Per-Protocol Population. Only those participants with PET data available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/cm^3
Arm/Group | Placebo | GSK3008348 1000 mcg
Number analyzed (Participants) | 2 | 5
mL/cm^3
  Baseline, n=2,5 | 1.664 (19.67) | 1.503 (37.32)
  24 hours post-dose PET scan 2, n=1,3: number analyzed (Participants) | 1 | 3
  24 hours post-dose PET scan 2, n=1,3 | 1.530 (NA) — NA indicates that geometric coefficient of variation was not calculated as there was only one data point. | 1.474 (24.43)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from Day 1 up to 62 days
Description: Intent-to-Treat population was used to assess AEs and SAEs.
Arm/Group | Placebo | GSK3008348 1000 mcg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 1/3 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | GSK3008348 1000 mcg (N=5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT03069989/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT03069989/SAP_001.pdf